CLINICAL TRIAL: NCT00889759
Title: The Role of Addition of High Resolution-CT in Outbreak Investigation of Tuberculosis
Brief Title: The Role of High Resolution-Computed Tomography (CT) in Tuberculosis (TB) Outbreak Investigation
Status: Completed | Type: Observational
Sponsor: Armed Forces Capital Hospital, Republic of Korea (Other Government)
Responsible Party: Sei Won Lee/Division chief of pulmonology, Armed Forces Capital Hospital
Other Study IDs: TBoutbreak
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Outbreaks
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the role of high-resolution computed tomography of the chest (HRCT) in the investigation of an outbreak of TB that developed in the South Korean army.

DETAILED DESCRIPTION:
Outbreak investigation including tuberculin skin test (TST), QuantiFERON® TB Gold In-Tube (QFT), and simple chest radiography (CXR) will be performed. For participants with any abnormal findings in these tests, HRCT will be carried out. Active pulmonary TB is diagnosed based on sputum studies or HRCT findings. In addition, participants with positive results both in TST and QTF will be treated as having a latent TB infection (LTBI). TST and QTF were repeated in participants with positive result in one of these tests. CXR will be repeated in all participants at 3 and 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All soldiers who assigned to the military battery where a tuberculosis outbreak occurred

Exclusion Criteria:

* Soldiers who could not complete study

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A military unit in South Korean Army
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital

REFERENCES:
- [Derived] Lee SW, Jang YS, Park CM, Kang HY, Koh WJ, Yim JJ, Jeon K. The role of chest CT scanning in TB outbreak investigation. Chest. 2010 May;137(5):1057-64. doi: 10.1378/chest.09-1513. Epub 2009 Oct 31. PMID 19880906